CLINICAL TRIAL: NCT04850742
Title: Feasibility of Tracheobronchial Reconstruction Using Bioengineered Aortic Matrices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201812035DINC
Record Dates: First submitted 2021-04-18; First posted 2021-04-20 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Trachea Diseases; Tracheal Stenosis; Lung Cancer; Tuberculosis; Tracheitis; Airway Disease
Keywords: tracheal reconstruction; bronchial reconstruction; cryopreserved aorta
MeSH Terms: conditions — Tracheal Diseases; Tracheal Stenosis; Lung Neoplasms; Tuberculosis; Tracheitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryopreserved aorta (Experimental): After resection of a segment of tracheal or bronchial lesion, reconstruct the airway with cryopreserved aortic allograft.
  Interventions: Procedure: Cryopreserved aorta

INTERVENTIONS:
Procedure: Cryopreserved aorta — After resection of the tracheal or bronchial lesion with standard surgical techniques, the airway gap is reconstructed with a segment of human cryopreserved (-80 celsius degree) aortic allograft, which was not matched by the ABO and leukocyte antigen systems. The anastomosis is performed with standard technique for airway anastomosis. An Ultraflex covered tracheobronchial stent is inserted to prevent collapse for the aortic graft.

SUMMARY:
We used a segment of cryopreserved aorta as a graft for reconstruction for long segment tracheobronchial lesion in human.

ELIGIBILITY:
Inclusion criteria:

* Patients with advanced benign or malignant lesions involving trachea or bronchi, and has failed conventional treatment.
* Patients with proximal pulmonary tumors that require surgical resection and has involved proximal airways which is indicated for a pneumonectomy, sleeve lobectomy, or carina resection.

Exclusion criteria:

* Less than 20-year-old
* Unable to obtain informed consent.
* Pulmonary tumors that can be treated with standard lobectomy.
* Unresectable locally advanced malignant tumors
* Malignant tumors with contralateral lymph nodes involvement.
* Malignant tumors with distal metastases; except for simple resectable brain metastasis.
* Tracheal lesions which can be treated with standard resection and direct anastomosis.
* Allergic to iodine
* Unable to tolerate standard lobectomy
* Has human immunodeficiency virus infection
* Tracheal stenosis at proximal 2 cm on upper trachea

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
90-day mortality | 90 days
  The rate of death at 90 days.

SECONDARY OUTCOMES:
90-day morbidity | 90 days
  The occurrence of complication including 1) anastomotic leakage, 2) pneumonia, 3) difficult weaning, 4) airway obstruction by granulation tissue, 5) stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shing Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinod E, Seguin A, Pfeuty K, Fornes P, Kambouchner M, Azorin JF, Carpentier AF. Long-term evaluation of the replacement of the trachea with an autologous aortic graft. Ann Thorac Surg. 2003 May;75(5):1572-8; discussion 1578. doi: 10.1016/s0003-4975(03)00120-6. PMID 12735581
- [Background] Martinod E, Seguin A, Holder-Espinasse M, Kambouchner M, Duterque-Coquillaud M, Azorin JF, Carpentier AF. Tracheal regeneration following tracheal replacement with an allogenic aorta. Ann Thorac Surg. 2005 Mar;79(3):942-8; discussion 949. doi: 10.1016/j.athoracsur.2004.08.035. PMID 15734409
- [Background] Seguin A, Radu D, Holder-Espinasse M, Bruneval P, Fialaire-Legendre A, Duterque-Coquillaud M, Carpentier A, Martinod E. Tracheal replacement with cryopreserved, decellularized, or glutaraldehyde-treated aortic allografts. Ann Thorac Surg. 2009 Mar;87(3):861-7. doi: 10.1016/j.athoracsur.2008.11.038. PMID 19231406
- [Background] Martinod E, Chouahnia K, Radu DM, Joudiou P, Uzunhan Y, Bensidhoum M, Santos Portela AM, Guiraudet P, Peretti M, Destable MD, Solis A, Benachi S, Fialaire-Legendre A, Rouard H, Collon T, Piquet J, Leroy S, Venissac N, Santini J, Tresallet C, Dutau H, Sebbane G, Cohen Y, Beloucif S, d'Audiffret AC, Petite H, Valeyre D, Carpentier A, Vicaut E. Feasibility of Bioengineered Tracheal and Bronchial Reconstruction Using Stented Aortic Matrices. JAMA. 2018 Jun 5;319(21):2212-2222. doi: 10.1001/jama.2018.4653. PMID 29800033
- [Background] Martinod E, Paquet J, Dutau H, Radu DM, Bensidhoum M, Abad S, Uzunhan Y, Vicaut E, Petite H. In Vivo Tissue Engineering of Human Airways. Ann Thorac Surg. 2017 May;103(5):1631-1640. doi: 10.1016/j.athoracsur.2016.11.027. Epub 2017 Jan 18. PMID 28109571